CLINICAL TRIAL: NCT04129008
Title: Effect of Indobufen Versus Aspirin on Gastric Acid Secretion and Gastroesophageal Reflux in Patients With Coronary Heart Disease and Gastroesophageal Reflux Disease Undergoing Dual Antiplatelet Therapy: a Prospective, Randomized, Double-blind, Double-dummy, Positive Drug Parallel Control Clinical Trials
Brief Title: GaStroEsophageal effeCt of indobUfen Versus aspiRin in Patients Undergoing Dual antiplatElet Therapy
Acronym: SECURE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Emergency & Critical Care Center, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019026
Record Dates: First submitted 2019-10-08; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease; Gastroesophageal Reflux Disease
Keywords: coronary heart disease; gastroesophageal reflux disease; indobufen; aspirin
MeSH Terms: conditions — Coronary Artery Disease; Gastroesophageal Reflux; Coronary Disease | interventions — indobufen; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indobufen (Experimental)
  Interventions: Drug: Indobufen and aspirin mimetic
- Aspirin (Active Comparator)
  Interventions: Drug: Aspirin and indobufen mimetic

INTERVENTIONS:
Drug: Indobufen and aspirin mimetic — Day 1 to 84±7: The first time: indobufen 100mg + aspirin mimetic; The second time: indobufen 100mg
  Arms: Indobufen
Drug: Aspirin and indobufen mimetic — Day 1 to 84±7: The first time : aspirin 100mg+ indobufen mimetic; The second time: indobufen mimetic
  Arms: Aspirin

SUMMARY:
The dual antiplatelet therapy based on aspirin plays an important role in the treatment of patients with coronary heart disease. Although aspirin is widely used and effective, it has many limitations in the long-term including increased risk of bleeding. In patients with coronary heart disease and gastroesophageal reflux disease, the symptoms of gastroesophageal reflux are usually aggravated after the application of aspirin. As an antiplatelet drug, indobufen can reversibly and selectively inhibit platelet cyclooxygenase-1 (COX-1), thereby blocking the synthesis of thromboxane B2 (TXB2) and exerting its antiplatelet effect, and it does not affect the production of prostaglandins and endothelial prostacyclins in gastrointestinal mucosa. It has less gastrointestinal injury and lower risk of bleeding. This project is to study the effects of indobufen or aspirin on gastric acid secretion and gastroesophageal reflux in patients with coronary heart disease and gastroesophageal reflux disease treated with dual antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Patients with stable and unstable angina pectoris receiving dual antiplatelet therapy (combined with clopidogrel)
* Coronary angiography indicating ≥50% stenosis in >2.0 mm vessels
* Gastroesophageal Reflux Disease Diagnostic Questionnaire Score (≥8)
* Signed informed consent

Exclusion Criteria:

* Acute myocardial infarction within 1 month before admission
* Patients undergoing treatment related to gastroesophageal reflux disease (e.g. proton pump inhibitors, etc.)
* Patients receiving other antiplatelet drugs (such as cilostazol) and oral anticoagulants
* Patients with cardiogenic shock (systolic blood pressure <90 mmHg and/or diastolic blood pressure <60 mmHg), severe heart failure (killip grade ≥3), hepatic insufficiency (AST/ALT more than twice the upper limit of normal value caused by non-cardiac diseases), prior stroke and renal dysfunction (GFR <60 ml/min)
* Those with active hemorrhage, hemorrhagic diseases or tendency to bleeding, especially those with a history of cerebral hemorrhage
* People who are known to be intolerant or allergic to aspirin, indobufen or clopidogrel
* Patients with malignant tumors or with life expectancy <2 years
* Pregnant women, lactating women, women of childbearing age who do not take effective contraceptive measures, or those who plan to conceive during the trial, or those who have positive results of HCG examination before the trial
* Those who have participated in other clinical trials or are currently participating in other clinical trials within one month before the trial
* According to the judgement of the researchers, patients could not complete the study or comply with the requirements of the study (e.g. memory or behavioral disorders, mental disorders, alcohol dependence, prior defaults)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-10-17 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage time of intragastric pH<4.0 during 24-hour intragastric pH monitoring | 2 weeks±4 days
  This parameter will be detected by 24-hour intragastric pH monitoring (Medical Measurement Systems, Netherlands)

SECONDARY OUTCOMES:
Median value of intragastric pH during 24-hour intragastric pH monitoring | 2 weeks±4 days
  This parameter will be detected by 24-hour intragastric pH monitoring (Medical Measurement Systems, Netherlands)
Frequency of indigestion occurrence | 2 weeks ±4 days, 12 weeks±7 days
Rate of bleeding events (BARC criteria) | 2 weeks ±4 days, 12 weeks±7 days
Gastroesophageal reflux disease questionnaire score (GerdQ score) | 2 weeks ±4 days, 12 weeks±7 days
  Min 0, max 18, and higher scores mean a worse outcome
AA-induced platelet inhibition rate (TEG method) | 2 weeks ±4 days
ADP-induced platelet inhibition rate (TEG method) | 2 weeks ±4 days
DeMeester score | 2 weeks ±4 days
  Min 0, no upper limit, and higher scores mean a worse outcome

OTHER OUTCOMES:
AA-induced platelet inhibition rate (LTA method) | 2 weeks±4 days
ADP-induced platelet inhibition rate (LTA method) | 2 weeks±4 days
Rate of major adverse cardiovascular event (MACE, including all-cause death, non-fatal myocardial infarction, ischemic stroke, ischemia-driven revascularization, or rehospitalization for heart failure) | 2 weeks±4 days, 12 weeks±7days
Rate of single endpoint of cardiovascular events, including cardiovascular death, non-fatal myocardial infarction, ischemic stroke, ischemic-driven revascularization, rehospitalization for heart failure, and all-cause death | 2 weeks±4 days, 12 weeks±7days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China